CLINICAL TRIAL: NCT02650271
Title: Adjuvant Entecavir or Tenofovir for Hepatitis B Virus Related Hepatocellular Carcinoma After Curative Hepatic Resection
Brief Title: Adjuvant Entecavir or Tenofovir for Postoperative HBV-HCC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Guangxi Medical University (Other)
Responsible Party: Principal Investigator, Jian-Hong Zhong, Director, Guangxi Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AEVT-HCC
Record Dates: First submitted 2016-01-05; First posted 2016-01-08 (Estimated); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Hepatocellular Carcinoma
Keywords: adjuvant; entecavir; hepatocellular carcinoma; hepatic resection
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — entecavir; Tenofovir

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Entecavir (Experimental): Patients will be received entecavir (10 mg/d) after 3 days of liver resection.
  Interventions: Drug: Entecavir
- Tenofovir (Active Comparator): Patients will be received tenofovir (1#/d) after 3 days of liver resection.
  Interventions: Drug: Tenofovir

INTERVENTIONS:
Drug: Entecavir — Patients will be received entecavir (10 mg/d) before liver resection.
  Other Names: ETV
  Arms: Entecavir
Drug: Tenofovir — Patients will be received tenofovir before liver resection.
  Arms: Tenofovir

SUMMARY:
This study aims to compare the effect of antiviral therapy with entecavir or tenofovir for hepatitis B virus-related hepatocellular carcinoma after radical hepatectomy. Included patients will randomly divide into two groups.

DETAILED DESCRIPTION:
Hepatocellular carcinoma (HCC) is associated with a poor prognosis, and its incidence has increased dramatically in many countries. Hepatectomy is a radical therapy for early-stage HCC. However, even after radical resection, the prognosis for HCC patients remains discouraging because of the high recurrence rate and frequent incidence of intrahepatic metastasis. Therefore, preventing HCC recurrence is very important.

Hepatitis B virus (HBV) infection is the major risk factor for HCC development in China. Some retrospective studies have shown that tenofovir or entecavir treatment for HBV-related HCC patients can effectively reduce the HCC recurrence rate and increase the survival rate after hepatectomy. However, which drug has more efficacy has not been addressed.

ELIGIBILITY:
Inclusion Criteria:

* Underwent hepatic resection.
* Diagnosis of HCC was confirmed by postoperative histopathology.
* Positive of HBsAg, HBeAg, or HBV DNA.
* Child-Pugh A or B liver function.

Exclusion Criteria:

* Anti-HCV(+)
* Diagnosis of HCC was not confirmed by postoperative histopathology of surgical samples after surgery.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2021-02-02 (Actual); Primary Completion 2023-12-25 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
overall survival | 1-year

SECONDARY OUTCOMES:
Recurrence rate | 1-year

OTHER OUTCOMES:
Perioperative reactivation of hepatitis B virus replication | 1-month

CONTACTS AND LOCATIONS:
Overall Officials: Le-Qun Li, MD, Study Chair — Guangxi Medical University Cancer Hospital
Locations (1):
- Department of Hepatobilliary Surgery, Affiliated Tumor of Guangxi University, Nanning, Guangxi, China

REFERENCES:
- [Background] Ke Y, Ma L, You XM, Huang SX, Liang YR, Xiang BD, Li LQ, Zhong JH. Antiviral therapy for hepatitis B virus-related hepatocellular carcinoma after radical hepatectomy. Cancer Biol Med. 2013 Sep;10(3):158-64. doi: 10.7497/j.issn.2095-3941.2013.03.006. PMID 24379991
- [Background] Kim SU, Seo YS, Lee HA, Kim MN, Lee YR, Lee HW, Park JY, Kim DY, Ahn SH, Han KH, Hwang SG, Rim KS, Um SH, Tak WY, Kweon YO, Kim BK, Park SY. A multicenter study of entecavir vs. tenofovir on prognosis of treatment-naive chronic hepatitis B in South Korea. J Hepatol. 2019 Sep;71(3):456-464. doi: 10.1016/j.jhep.2019.03.028. Epub 2019 Apr 6. PMID 30959156
- [Background] Teng YX, Li MJ, Xiang BD, Zhong JH. Tenofovir may be superior to entecavir for preventing hepatocellular carcinoma and mortality in individuals chronically infected with HBV: a meta-analysis. Gut. 2020 Oct;69(10):1900-1902. doi: 10.1136/gutjnl-2019-320326. Epub 2019 Dec 16. No abstract available. PMID 31843789
- [Background] Yuan BH, Li RH, Huo RR, Li MJ, Papatheodoridis G, Zhong JH. Lower risk of hepatocellular carcinoma with tenofovir than entecavir treatment in subsets of chronic hepatitis B patients: an updated meta-analysis. J Gastroenterol Hepatol. 2022 May;37(5):782-794. doi: 10.1111/jgh.15783. Epub 2022 Feb 7. PMID 35080052
- [Background] Pan LX, Wang YY, Li ZH, Luo JX, Wu KJ, Liu ZX, Wu PS, Chen K, Ma L, Fan XH, Zhong JH. Entecavir versus tenofovir for prevention of hepatitis B virus-associated hepatocellular carcinoma after curative resection: study protocol for a randomized, open-label trial. Trials. 2024 Jan 5;25(1):25. doi: 10.1186/s13063-023-07742-x. PMID 38183137